CLINICAL TRIAL: NCT01812941
Title: Evaluation of Mitochondrial Dysfunction in Severe Burn and Trauma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Alabama (Other)
Responsible Party: Principal Investigator, Jon Simmons, Principal investigator, University of South Alabama
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 11-212
Record Dates: First submitted 2013-03-13; First posted 2013-03-18 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Burns; Trauma
Keywords: burns; trauma
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Burn: blood collection (Other): Procedure: Blood draws as the intervention.
  Interventions: Other: Burn: blood collection
- trauma: blood collection (Other): blood to be collected at different time intervals. Blood draw as the intervention
  Interventions: Other: trauma: blood collection
- healthy volunteers: blood collection (Other): Blood draws as the intervention
  Interventions: Other: healthy volunteers: blood collection

INTERVENTIONS:
Other: trauma: blood collection — Blood samples collected at certain timepoints. Time points for burn/trauma subjects: Day0,Day1,Day2,and Day6 and Day7.
  Arms: trauma: blood collection
Other: healthy volunteers: blood collection — blood collected at designated time intervals
  Arms: healthy volunteers: blood collection
Other: Burn: blood collection — blood collected at designated time intervals
  Arms: Burn: blood collection

SUMMARY:
The purpose of this project is to evaluate the level of mitochondrial dysfunction several patient populations: Burn, trauma, and control group of healthy volunteers.

Study hypothesis: Increased plasma concentrations of a newly discovered inflammatory mediated, called mtDNA DAMPS associated with the occurrence of multi-organ dysfunction syndrome in severly injured patients.

As the severity of a burn injury or trauma injury increase, so will systemic mitochondrial dysfunction.

DETAILED DESCRIPTION:
Increased plasma concentrations of a newly discovered inflammatory mediated, called mtDNA DAMPS associated with the occurrence of multi-organ dysfunction syndrome in severly injured patients.

A normal healthy sub-population will be used as a control.

ELIGIBILITY:
Inclusion Criteria:

* Burn injury must be less than 24 hours old at time of initial sampling
* Burn must be 2nd or 3rd degree and at least 10% TBSA
* ISS (injury severity score) > 15

Exclusion Criteria:

* Burn injury/trauma injury > than 24hours old at time of initial sampling
* Burn < 10% total body surface area.
* Evidence of active infection on admission in the burn subjects.
* < 19 years of age and > 70 years

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-09; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Plasma mtDNA DAMPs concentration | approximately 1 year to assess outcome measure
  Plasma mtDNA DAMPs concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jon Simmons, MD, Principal Investigator — University of South Alabama, Department of Surgery
Locations (1):
- University of South Alabama Medical Center, Mobile, Alabama, United States

REFERENCES:
- [Derived] Simmons JD, Lee YL, Mulekar S, Kuck JL, Brevard SB, Gonzalez RP, Gillespie MN, Richards WO. Elevated levels of plasma mitochondrial DNA DAMPs are linked to clinical outcome in severely injured human subjects. Ann Surg. 2013 Oct;258(4):591-6; discussion 596-8. doi: 10.1097/SLA.0b013e3182a4ea46. PMID 23979273